CLINICAL TRIAL: NCT01201005
Title: B VITAMIN STATUS IN PREMATURE AND SMALL FOR GESTATIONAL AGE INFANTS
Brief Title: B Vitamin Status in Premature and Small for Gestational Age(SGA) Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Haukeland University Hospital (Other)
Responsible Party: Anne-Lise Bjørke Monsen, Haukeland University Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: REK-Vest 104.08
Record Dates: First submitted 2010-09-12; First posted 2010-09-14 (Estimated); Last update posted 2010-09-14 (Estimated); Status verified 2010-09

CONDITIONS: Biochemical Cobalamin Status; Motor Neurodevelopment
MeSH Terms: interventions — Hydroxocobalamin; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Hydroxycobalamin (Active Comparator): Hydroxycobalamin 400 µg (Vitamin B12 depot, Nycomed Pharma) is given as a singel intramuscular injection.
  The syringe is covered so it is impossible to see whether it contains any substance
  Interventions: Dietary Supplement: Hydroxycobalamin
- needle injection (Sham Comparator): The controls receive an intramuscular "injection": which is merely an introduction of the needle into the muscle whithout any injection. The syringe is covered so it is not possible to see whether the syringe contains any substance
  Interventions: Dietary Supplement: Sham injection

INTERVENTIONS:
Dietary Supplement: Hydroxycobalamin — Hydroxycobalamin 400 µg (Vitamin B12 depot, Nycomed Pharma ) is given as a single intramuscular injection
  Arms: Hydroxycobalamin
Dietary Supplement: Sham injection — needle injection without any substance given
  Arms: needle injection

SUMMARY:
Premature birth and low birth weight implies insufficient intrauterine growth and fetal malnutrition. During the first months of life where the infant is breastfed, the low stores aquired during fetal life, may cause specific B vitamin deficiencies. In this study infants with a birth weight below 3000 g will be studied at 6 weeks, 4 and 6 months. At 6 months infants with biochemical signs of impaired cobalamin status (i.e.: tHcy > 97.5 percentile for cobalamin treated infants, i.e.: tHcy>6.5 µM/L) will be randomised to cobalamin treatment or placebo. At 7 months the investigators will evaluate the effect of cobalamin or placebo treatment according to infant biochemical status and neurodevelopment.

Study hypothesis: Cobalamin treatment given to infants with biochemical cobalamin deficiency will normalize biochemical status and cause improved motor neurodevelopment.

ELIGIBILITY:
Inclusion Criteria:

* Birthweight < 3000 grams
* Age 6 months (+/- 0.5 months)
* Plasma total homocysteine > 6.5 umol/L

Exclusion Criteria:

* Plasma total homocysteine < 6.5 umol/L

Ages: 5 Months to 7 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 80 (Actual)
Dates: Start 2009-07; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Changes in biochemical status and neurodevelopment | 4 weeks
  Bloodsamples for analysis of B vitamin status are drawn before intervention and after 4 weeks Neurological evaluation (AIMS test) of the infants is done before intervention and after 4 weeks

SECONDARY OUTCOMES:
Maternal evaluation of changes in infant behaviour/development | 4 weeks
  Maternal evaluation of changes in infant behaviour will be tested by using a maternal questionnaire, Ages and Stages (ASQ), a highly rated child screening and monitoring system, before and after intervention

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Norway

REFERENCES:
- [Background] Bjorke-Monsen AL, Torsvik I, Saetran H, Markestad T, Ueland PM. Common metabolic profile in infants indicating impaired cobalamin status responds to cobalamin supplementation. Pediatrics. 2008 Jul;122(1):83-91. doi: 10.1542/peds.2007-2716. PMID 18595990
- [Derived] Torsvik IK, Ueland PM, Markestad T, Midttun O, Bjorke Monsen AL. Motor development related to duration of exclusive breastfeeding, B vitamin status and B12 supplementation in infants with a birth weight between 2000-3000 g, results from a randomized intervention trial. BMC Pediatr. 2015 Dec 18;15:218. doi: 10.1186/s12887-015-0533-2. PMID 26678525
- [Derived] Torsvik IK, Markestad T, Ueland PM, Nilsen RM, Midttun O, Bjorke Monsen AL. Evaluating iron status and the risk of anemia in young infants using erythrocyte parameters. Pediatr Res. 2013 Feb;73(2):214-20. doi: 10.1038/pr.2012.162. Epub 2012 Nov 20. PMID 23168578